CLINICAL TRIAL: NCT04093297
Title: Flexible Band Versus Rigid Ring Annuloplasty for the Correction of Tricuspid
Brief Title: Band Versus Ring for Tricuspid Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Staff of Department of Cardiothoracic Surgery, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JPH2019
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ring (Active Comparator): Patients in Group Ring will undergo tricuspid rigid ring annuloplasty
  Interventions: Procedure: Tricuspid Annuloplasty
- Group Band (Active Comparator): Patients in Group Band will undergo flexible band annuloplasty
  Interventions: Procedure: Tricuspid Annuloplasty

INTERVENTIONS:
Procedure: Tricuspid Annuloplasty — Patients will undergo repair of tricuspid regurgitation

SUMMARY:
Tricuspid regurgitation is common in patients with heart valve disease, both flexible band and rigid ring annuloplasty can correct this anomaly. However, there is no data to address which one can bring more benefits to these patients with combined heart valve disease. This study aims to prospectively compare the efficacy and long term outcomes of flexible band versus rigid ring annuloplasty for the correction of tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject must be 18 years and 80 years at time of consent and must not be a member of a vulnerable population.
* 2. Subject or a legally authorized representative (where allowed per local regulations) must provide written informed consent prior to any trial related procedure.
* 3. Subjects with moderate or greater tricuspid regurgitation determined by the assessment of a qualifying transthoracic echocardiogram (TTE) and/or transesophageal echocardiogram (TEE).
* 4. Subjects with moderate tricuspid regurgitation will only be included in the trial if moderate tricuspid regurgitation is accompanied by a tricuspid annular diameter of ≥ 40mm as measured by echocardiography.
* 5. Isolated functional symptomatic tricuspid regurgitation of moderate to severe or greater, with annular dilatation of ≥ 40mm;
* 6. Requirement for concomitant left heart valve surgery;
* 7. Requirement for concomitant coronary artery surgery;
* 8. Requirement for concomitant atrial fibrillation surgery;
* 9. Available and able to return to the study site for post-procedural follow-up examination;

Exclusion Criteria:

* 1. Patient unable or unwilling to provide informed consent;
* 2. Subjects with mild tricuspid regurgitation;
* 3. Emergency surgery;
* 4. Prior tricuspid valve leaflet surgery or any currently implanted prosthetic tricuspid valve, or any prior transcatheter tricuspid valve procedure;
* 5. Subjects with percutaneous coronary intervention within prior 30 days prior to enrollment;
* 6. Subjects with presence of any known life threatening (non-cardiac major or progressive disease), non-cardiac disease that will limit the subject's life expectancy to less than one year;
* 7. Subjects with permanent or temporary pacemaker implantation;
* 8. Subjects with severe, irreversible pulmonary hypertension in the judgment of the investigator;
* 9. History of mitral/tricuspid endocarditis within the last 12 months;
* 10. Subjects with contraindication or known allergy to device's components, aspirin, anti-coagulation therapy or contrast media that cannot be adequately premeditated;
* 11. Subjects with bleeding or coagulation disorders (e.g. active peptic ulcer or active gastrointestinal bleeding);
* 12. Female patient is pregnant (urine HCG test result positive) or lactating;
* 13. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint;
* 14. Subjects with left ventricular ejection fraction (LVEF)≤20%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of reoperation for tricuspid regurgitation, progression of tricuspid regurgitation by two grades from baseline or the presence of severe tricuspid regurgitation, or death. | at follow-up of 5 years
  Improvement in tricuspid regurgitation: refers to Mild or No tricuspid regurgitation Tricuspid regurgitation is graded as mild, moderate, and severe based on regurgitant jet area

SECONDARY OUTCOMES:
Mortality | up to 3 months of intervention
  Mortality: Mortality within hospital stay or 1 month postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Veen KM, Etnel JRG, Quanjel TJM, Mokhles MM, Huygens SA, Rasheed M, Oei FBS, Ten Cate FJ, Bogers AJJC, Takkenberg JJM. Outcomes after surgery for functional tricuspid regurgitation: a systematic review and meta-analysis. Eur Heart J Qual Care Clin Outcomes. 2020 Jan 1;6(1):10-18. doi: 10.1093/ehjqcco/qcz032. PMID 31287501